CLINICAL TRIAL: NCT03019913
Title: Evaluation of Bedside Methods to Measure Muscularity in Critically Ill Patients: A Prospective Observational Study
Brief Title: Evaluation of Bedside Methods to Measure Muscularity in Critically Ill Patients
Status: Completed | Type: Observational
Sponsor: La Trobe University (Other)
Collaborators: The Alfred (Other)
Responsible Party: Principal Investigator, Kate Lambell, PhD candidate, Dietitian, La Trobe University
Other Study IDs: 523/16
Record Dates: First submitted 2017-01-11; First posted 2017-01-13 (Estimated); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Critical Illness
Keywords: Skeletal muscle
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Observational cohort — Evaluation of bedside methods to measure muscularity in critically ill patients

SUMMARY:
Muscle wasting is a significant problem in critically ill patients, with reported losses of a half to three percent per day over the first ten days (for an average 70kg person this equates to 3 to 20kg of muscle loss). Low skeletal muscle mass at admission to the intensive care unit (ICU) and the loss of lean tissue have been associated with negative clinical outcomes, including increased incidence of infections, length of stay, mortality and muscle weakness. It is therefore crucial that technology is utilised to: 1) identify ICU patients with low muscularity on admission, 2) to help understand the factors impacting muscle loss and to 3) assess the effectiveness of interventions aimed at maintaining skeletal muscle mass in this population.

The measurement of lean body mass in patients admitted to the ICU is challenging however, due to the large fluid shifts that occur in this population and logistical issues in moving patients to specialised machinery for body composition analysis. Currently, there is no validated method for accurately assessing a patient's muscle mass at the bedside in the intensive care setting. It is therefore important to investigate the accuracy, feasibility and reliability of bedside methods such as subjective physical assessment of muscle mass, mid arm muscle circumference, ultrasound and bioimpedance analysis to assess muscularity in this population who are primarily bedbound. In order to do this, a critical comparison is required between these methods and muscularity assessed by a "reference" body composition method, such computed tomography (CT) image analysis. Briefly, quantification of skeletal muscle at the abdomen area utilising abdominal CT images has been shown to be highly representative of whole body skeletal muscle volume.

We wish to conduct a pilot, feasibility study (n= 50), which will recruit patients who have a CT scan (containing abdomen area), performed for clinical purposes. Our primary aim will be to investigate whether muscularity assessed with non-invasive bedside methods (ultrasound, bioimpedance analysis, SGA physical assessment, mid arm muscle circumference) are correlated with skeletal muscle mass quantified by a "reference method" (CT image analysis).

DETAILED DESCRIPTION:
Aim Our primary aim is to investigate whether muscularity assessed via bedside ultrasound is correlated with a reference method for estimating whole body skeletal muscle mass (CT image analysis) in the first few days of critical illness.

Our secondary aims are

* To investigate whether muscularity assessed via other bedside methods (bioimpedance spectroscopy, subjective physical assessment and mid arm muscle circumference) are correlated with a reference method for estimating whole body skeletal muscle mass (CT image analysis) in critically ill patients.
* To better understand the association between measured resting energy expenditure and muscularity in the critically ill.
* To observe changes in skeletal muscle mass (in a sub set of patients who have two CT scans) and the impact various factors, including energy and protein delivery has on these changes.

ELIGIBILITY:
Inclusion Criteria:

* Have had a CT scan of the L3 vertebra performed for clinical reasons ≤24 hours before or ≤72 hours after ICU admission

Exclusion Criteria:

* CT scan performed >48hrs ago
* Death is imminent or deemed highly likely in the next 96 hours
* Are known to be pregnant
* Treating clinician does not believe the study to be in the best interest of the patient
* It is not possible to image two or more muscle groups via ultrasound (i.e. due to trauma, burns, wounds)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill adults
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-01; Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Mean skeletal muscle mass measured by CT scan analysis at L3 area (cm2) | CT performed for clinical reasons ≤24 hours before or ≤72 hours after ICU admission
Mean skeletal muscle mass measured by ultrasound (muscle thickness at each site, cm and rectus femoris CSA, cm2) | <48 hours after CT scan containing L3 area

SECONDARY OUTCOMES:
Fat free mass (kg), phase angle and impedance ratio measured by bioimpedance spectroscopy | <48 hours after CT scan containing L3 area
Subjective assessment of muscle and fat wasting via SGA (normal, mild-moderate or severe) | <48 hours after CT scan containing L3 area
Mid arm muscle circumference (cm) | <48 hours after CT scan containing L3 area
Mean skeletal muscle mass measured by CT scan analysis at femoral area (cm2) | CT performed for clinical reasons ≤24 hours before or ≤72 hours after ICU admission
Measured resting energy expenditure (kilojoules) | <48 hours after CT scan containing L3 area
Intramuscular, subcutaneous and visceral adipose tissue CSA at L3 area (cm2) | CT performed for clinical reasons ≤24 hours before or ≤72 hours after ICU admission

CONTACTS AND LOCATIONS:
Overall Officials: Kate Lambell, MNutrDiet, Principal Investigator — La Trobe University and Alfred Health
Locations (1):
- The Alfred Hospital, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lambell KJ, Tierney AC, Wang JC, Nanjayya V, Forsyth A, Goh GS, Vicendese D, Ridley EJ, Parry SM, Mourtzakis M, King SJ. Comparison of Ultrasound-Derived Muscle Thickness With Computed Tomography Muscle Cross-Sectional Area on Admission to the Intensive Care Unit: A Pilot Cross-Sectional Study. JPEN J Parenter Enteral Nutr. 2021 Jan;45(1):136-145. doi: 10.1002/jpen.1822. Epub 2020 Apr 15. PMID 32291773